CLINICAL TRIAL: NCT04825158
Title: Study of the Role of Hemostasis in Perioperative Anaphylaxis
Acronym: HEMOCANOPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8030
Record Dates: First submitted 2021-01-21; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hemoptysis; Perioperative Complication; Anaphylaxis
MeSH Terms: conditions — Hemoptysis; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Whole blood
  * Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anaphylaxis is a severe and life-threatening complication during the perioperative period. Perioperative anaphylaxis is still associated with a significant mortality despite quick and efficient management using epinephrine, the mainstay of acute treatment. Experimental data and few case reports are suggesting that hemostasis, and more precisely platelets, could play a role in anaphylaxis. Our main hypothesis is that activation of the hemostatic system contributes to the severity of the reaction

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, adult
* In the perioperative period
* In whom the diagnosis of anaphylactic shock is suggested
* Patient is giving his consent to participate in the study

Exclusion Criteria:

* Subject under legal protection
* Subject under guardianship or guardianship
* Anemia less than 7 g /dl at the time of inclusion

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will focus on any adult patient with a suspected diagnosis of perioperative anaphylactic shock
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2024-02-09 (Estimated)

PRIMARY OUTCOMES:
Platelet activation | As soon as possible after onset of anaphylaxis
  Measurement of: Plasmatic serotonin level, Plasmatic PF-4 level, P-selectin expression (MFI, %), Platelet count
Platelet activation | 1-2 hours after the onset of anaphylaxis
  Measurement of: Plasmatic serotonin level, Plasmatic PF-4 level, P-selectin expression (MFI, %), Platelet count
Platelet activation | 24 hours after the onset of anaphylaxis
  Measurement of: Plasmatic serotonin level, Plasmatic PF-4 level, P-selectin expression (MFI, %), Platelet count
Platelet activation | During the allergic workup (4-6 weeks after)
  Measurement of: Plasmatic serotonin level, Plasmatic PF-4 level, P-selectin expression (MFI, %), Platelet count